CLINICAL TRIAL: NCT03180970
Title: Different Lugol's Solution Concentration for Image Quality of Early Esophageal Squamous Neoplasia in Chromoendoscopy With Iodine Staining
Brief Title: Different Lugol's Solution Concentration for Image Quality of Esophageal Lesions in Chromoendoscopy With Iodine Staining
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Xiuli Zuo, director of Qilu Hospital, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2017SDU-QILU-G002
Record Dates: First submitted 2017-06-04; First posted 2017-06-08 (Actual); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Image Quality of Early Esophageal Squamous Neoplasia; Endoscopists'Subjective Assessments
MeSH Terms: interventions — Lugol's solution

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- group 1 (Experimental): This group patients were given dosages of 1.2% Lugol's solution for chromoendoscopy.
  Interventions: Drug: 1.2% Lugol's solution
- group 2 (Experimental): This group patients were given dosages of 1.0% Lugol's solution for chromoendoscopy.
  Interventions: Drug: 1.0% Lugol's solution
- group 3 (Experimental): This group patients were given dosages of 0.8% Lugol's solution for chromoendoscopy.
  Interventions: Drug: 0.8% Lugol's solution
- group 4 (Experimental): This group patients were given dosages of 0.6% Lugol's solution for chromoendoscopy.
  Interventions: Drug: 0.6% Lugol's solution
- group 5 (Experimental): This group patients were given dosages of 0.4% Lugol's solution for chromoendoscopy.
  Interventions: Drug: 0.4% Lugol's solution

INTERVENTIONS:
Drug: 1.2% Lugol's solution — 1.2% Lugol's solution will be sprayed on the lesion suspected early esophageal squamous neoplasia .Then the lesions will be treated with endoscopic submucosal dissection(ESD).
  Arms: group 1
Drug: 1.0% Lugol's solution — 1.0% Lugol's solution will be sprayed on the lesion suspected early esophageal squamous neoplasia .Then the lesions will be treated with endoscopic submucosal dissection(ESD).
  Arms: group 2
Drug: 0.8% Lugol's solution — 0.8% Lugol's solution will be sprayed on the lesion suspected early esophageal squamous neoplasia .Then the lesions will be treated with endoscopic submucosal dissection(ESD).
  Arms: group 3
Drug: 0.6% Lugol's solution — 0.6% Lugol's solution will be sprayed on the lesion suspected early esophageal squamous neoplasia .Then the lesions will be treated with endoscopic submucosal dissection(ESD).
  Arms: group 4
Drug: 0.4% Lugol's solution — 0.4% Lugol's solution will be sprayed on the lesion suspected early esophageal squamous neoplasia .Then the lesions will be treated with endoscopic submucosal dissection(ESD).
  Arms: group 5

SUMMARY:
The purpose of this study is to assess whether lower Lugol's solution concentration can perceive the same image quality of early esophageal squamous neoplasia.

DETAILED DESCRIPTION:
Chromoendoscopy using Lugol's solution is effective for the detection of early esophageal squamous neoplasia. However, this modality may cause severe chest pain and discomfort owing to mucosal irritation.

This study was to test whether a lower concentration of Lugol's solution can provide satisfied image quality of early esophageal squamous neoplasia and has lower mucosal irritation.

ELIGIBILITY:
Inclusion Criteria:

Patients with early esophageal squamous neoplasia who underwent endoscopic submucosal dissection.

Exclusion Criteria:

After esophageal surgery or endoscopic treatment ; Known esophageal radiotherapy or chemotherapy ; Esophageal stenosis; Acute bleeding; A known allergy to iodine; Coagulopathy (prothrombin time <50% of control, partial thromboplastin time >50 seconds); Having food retention; Severe hepatic ,renal, cardiovascular or metabolic dysfunction ; Being pregnant or lactating.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Image Quality of Esophageal Lesions | seven months
  Evaluated by Image J software (National Institutes of Health)

SECONDARY OUTCOMES:
Questionnaire of endoscopists' subjective assessments | intraoperative
  The picture will be rated for quality according to color contrast of esophageal lesions after iodine sprayed by the endoscopist performing the examination
Complete resection/R0 resection rate | 1 month
Mucosal change of the stomach in white-light endoscopy after Lugol's solution sprayed. | intraoperative
  The endoscopic findings of the greater curvature of the gastric body where the agent collected will be evaluated based on the following findings:fold thickening, exudates, ulcers, and hemorrhage.
The amount of Lugol's solution | intraoperative
Severe adverse events (allergic reactions, esophageal burns, spasms and even perforation) | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Zuo, PhD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital, Shandong University, Jinan, Shandong, China